CLINICAL TRIAL: NCT06531954
Title: Comparison Of Breathing Exercises and Auricular Vagus Nerve Stimulation Effects On Autonomic Nervous System Activity and Respiratory Functions In Healthy Adults
Brief Title: Breathing Exercises and Auricular Vagus Nerve Stimulation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, gulay karacaoglu, Doctor, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Nervusvagus
Record Dates: First submitted 2024-07-24; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Breathing Exercises; Auricular Vagus Nerve Stimulation; Autonomic Nervous System
Keywords: Breathing Exercises; Autonomic Nervous System; Pulse Rate Variability; Respiratory Functions; Auricular Vagus Nerve Stimulation
MeSH Terms: interventions — Vagus Nerve Stimulation; Breathing Exercises

STUDY DESIGN:
Intervention Model Description: Our study was conducted as a randomized prospective study. In both groups, the interventions were performed for ten sessions for two weeks, five days a week. In both groups, heart rate variability, heart rate, and blood tension were measured before and after each session, and the pulmonary function test was evaluated the day before and the day after the ten sessions of applications.
Who Masked: Participant
Masking Description: The 88 volunteer cases were divided into two groups by randomization. By randomization, according to the order of participation in the study, odd-numbered people (such as first, third, fifth) were included in the breathing exercises group (Group BE); even-numbered people (such as second, fourth, sixth) were included in the vagus nerve stimulation group (Group VNS). After randomization, 44 cases in Group BE and 44 cases in Group VNS were evaluated. All participants completed the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathing exercise group (BE) (Active Comparator): The content of breathing exercises was planned as thoracic expansion exercises. These exercises were applied to the lower, middle, and upper lobes in 3 sets of 3x10 (90 times breathing in one area) and lasted for an average of 20 minutes. These exercises were first taught by the physiotherapist and performed under her supervision. Participants were asked to inhale as deeply as possible into the relevant area, hold their breath for 3 seconds, and then slowly exhale the entire breath.
  Interventions: Behavioral: Breathing exercise
- Vagus nerve stimulation group (VNS) (Experimental): Vagus stimulation was applied bilaterally through the ear. taVNS was performed with the Vagustim device. The stimulation pulse width was 300 microseconds, the frequency was 10 Hz, and it was biphasic with a 20-minute duration. Electrodes were placed on the concha and tragus parts of the ear, and the current was increased through these electrodes until the participant felt pain. When the participant felt pain, the intensity was reduced to a comfortable sensation.
  Interventions: Device: Vagus nerve stimulation

INTERVENTIONS:
Device: Vagus nerve stimulation — Vagus nerve stimulation group: Vagus stimulation was applied bilaterally through the ear. taVNS was performed with the Vagustim device. The stimulation pulse width was 300 microseconds, the frequency was 10 Hz, and it was biphasic with a 20-minute duration. Electrodes were placed on the concha and tragus parts of the ear, and the current was increased through these electrodes until the participant felt pain.
  Arms: Vagus nerve stimulation group (VNS)
Behavioral: Breathing exercise — Breathing exercise group: The content of breathing exercises was planned as thoracic expansion exercises. These exercises were applied to the lower, middle, and upper lobes in 3 sets of 3x10 (90 times breathing in one area) and lasted for an average of 20 minutes. Participants were asked to inhale as deeply as possible into the relevant area, hold their breath for 3 seconds, and then slowly exhale the entire breath.
  Arms: Breathing exercise group (BE)

SUMMARY:
Introduction: Vagal modulation is achieved directly by transcutaneous auricular vagus nerve stimulation, whereas breathing exercises stimulate arterial baroreceptors. In this study, we aimed to compare these two methods, which have similar effects.

Methods: 88 healthy participants aged 18-35 were randomly divided into breathing exercises (Group BE) and vagus stimulation (Group VNS). Thoracic expansion exercise was performed in the BE group. In the VNS group, biphasic electrical stimulation was applied to both ears with a pulse width of 300 microseconds, frequency of 10 Hz, and 20 minutes. Pulmonary function tests were measured on the first and last day. Heart rate, systolic and diastolic blood pressure, RMSSD, PNN50, LF/HF, LF Power, and HF Power values were measured before and after each of the ten sessions for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals between the ages of 18 and 35,
* without orthopedic disability,
* without any chronic disease and regular medication use,
* who had not smoked for the last year,
* who had no problems in reading, writing, or comprehension were included in our study.

Exclusion Criteria:

* active or chronic respiratory diseases and communication problems because they may adversely affect pulmonary function testing

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2021-01-02 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Autonomic nervous system activity | pre-intervention, immediately after-intervention
  Autonomic measurements of each individual participating in the study before and after the intervention were performed with heart rate variability parameters. For this purpose, the Elite HRV device was used. The device has a finger sensor and an application compatible with the phone. Elite HRV application is a software that can synchronize with a personal monitor by collecting peak-to-peak intervals for instant analysis of pulse rate variability (PRV). In addition to all these assessments, blood pressure measurements of the participants were also evaluated using an Omron M2 electronic sphygmomanometer on the right arm.
Pulmonary Function. Forced expiratory volume in the first second (FEV1) | pre-intervention, immediately after-intervention
  Participants in both groups underwent pulmonary function test evaluation on the first and last day. Since the study was conducted in healthy individuals, it was deemed appropriate to look at the pulmonary function test before and after exertion to see possible changes. Medwelt SP10 spirometer was used for pulmonary function tests in our study. Each individual was measured in a sitting position using a separate mouthpiece.
Pulmonary Function. Forced vital capacity (FVC) | pre-intervention, immediately after-intervention
  Participants in both groups underwent pulmonary function test evaluation on the first and last day. Since the study was conducted in healthy individuals, it was deemed appropriate to look at the pulmonary function test before and after exertion to see possible changes. Medwelt SP10 spirometer was used for pulmonary function tests in our study. Each individual was measured in a sitting position using a separate mouthpiece.

CONTACTS AND LOCATIONS:
Locations (1):
- Mudanya University, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Our study was conducted as a randomized prospective study. In both groups, the interventions were performed for ten sessions for two weeks, five days a week. In both groups, heart rate variability, heart rate, and blood tension were measured before and after each session, and the pulmonary function test was evaluated the day before and the day after the ten sessions of applications. Since the study was conducted in healthy participants, pulmonary function tests were examined Before and after aerobic training to see possible changes. The training on the treadmill consisted of 5-minute warm-ups, 20 minutes of loading, and five 5-minute cool-down periods. Participants performed warm-up and cool-down periods at a treadmill speed of 4km/h. After determining the maximum heart rate according to the 220-age formula, the loading intensity was performed at 60% of this value [4]. Intergroup comparisons were made as a result of the evaluations in both groups.
Supporting Information: Study Protocol
Time Frame: a year
Access Criteria: nervus vagus stimulation

REFERENCES:
- [Result] Hatik SH, Arslan M, Demirbilek O, Ozden AV. The effect of transcutaneous auricular vagus nerve stimulation on cycling ergometry and recovery in healthy young individuals. Brain Behav. 2023 Dec;13(12):e3332. doi: 10.1002/brb3.3332. Epub 2023 Nov 16. PMID 37974551